CLINICAL TRIAL: NCT04272827
Title: Multicentre, Controlled, Randomized, Investigator-blinded Clinical Trial on Efficacy and Safety of Surgical Therapy of Lipedema Compared to Complex Physical Decongestive Therapy Alone (LIPLEG)
Brief Title: Evaluation Between Surgical Therapy of Lipedema Compared to Complex Physical Decongestive Therapy (CDT) Alone
Acronym: LIPLEG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hautklinik Darmstadt (Other)
Collaborators: The Clinical Trials Centre Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIPLEG-3806
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-03

CONDITIONS: Lipedema
Keywords: Lipedema; complex decongestive therapy(CDT); liposuction
MeSH Terms: conditions — Lipedema | interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: After a run in phase, randomization is performed in the intervention and control arm (2:1).
Who Masked: Outcomes Assessor
Masking Description: Random assignment of patients to one of the two treatment groups (experimental or controlled) is provided centrally via a 24/7 Internet service in ratio 2:1 (experimental: controlled) based on permuted blocks. The assignment is stratified to stage and centre.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): In the intervention group, patients will receive liposuction treatment (number of surgeries at the discretion of the attending study physician: a maximum of 4 surgical procedures, with a minimum of 5 and a maximum of 7 weeks between each surgery) with concomitant complex decongestive therapy (CDT), if necessary, to maintain surgical outcomes as required by the patient.
  Interventions: Procedure: Liposuction
- Control group (Other): After randomisation, the control group will be treated for 12 months with complex decongestive therapy (CDT) alone.
  After these 12 months, patients can opt for liposuction treatment if they continue to meet the inclusion and exclusion criteria.
  Interventions: Procedure: Liposuction

INTERVENTIONS:
Procedure: Liposuction — Liposuction treatment will be performed according to the study protocol using the "wet technique" depending on the amount of fat to be removed, if necessary in several sessions.

SUMMARY:
The purpose of this study is to determine whether surgical treatment of lipedema (stage I, II or III) using liposuction significantly improves leg pain compared to the use of complex decongestive therapy (CDT).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients that gave written informed consent will undergo a run-in phase of up to seven months for edema elimination and maintenance of results using complex decongestive therapy (CDT). Afterwards, patients will be assigned to one of the two treatment groups via internet randomization, provided that all inclusion and exclusion criteria continue to be met. Randomization will be 2:1 (intervention: control). In the intervention arm, patients will receive liposuction treatment (number of surgeries at the discretion of the treating study physician: a maximum of four surgical procedures, with a minimum of 5 and a maximum of 7 weeks between each surgery) with, if necessary, concomitant CDT to maintain the surgical results as required by the patient.

The primary endpoint (regarding pain in the legs in stages I, II or III) will be assessed after an observation period of 12 months after final liposuction surgery. This is followed by a further follow-up period for 24 months to observe and document the further course.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Female
3. Age ≥ 18 years
4. Confirmed lipedema of the legs in stage I, II or III
5. Average pain in the legs for the last four weeks ≥ 4 points on a numerical rating scale
6. Documentation of insufficient relief of symptoms by conservative measures
7. Willingness and ability to perform conservative measures according to the study protocol, during and, if necessary, after liposuction treatment
8. Full legal capacity

Exclusion Criteria:

1. Concurrent lipedema of the arms and legs, in which co-occurrence of lipedema in the arms affects the primary endpoint (i.e., average leg pain), at the discretion of the study investigator
2. Previous liposuctions
3. Diseases that may limit operability at the discretion of the study physician, e.g. cardiac diseases, coagulation disorders, metabolic diseases, infectious diseases (active), epilepsy; diseases requiring immunosuppression or anticoagulation with medication; allergies to medication accompanying surgery
4. Weight >120.0 kg
5. Medical conditions that affect adequate complex decongestive therapy (CDT) at the discretion of the study physician, e.g. heart failure (volume stress), lack of physical ability to wear compression stockings (e.g. joint disease, neurological deficits).
6. Primary obesity without disproportion and without evidence of lipedema
7. Secondary obesity
8. Fat distribution disorders of other genesis (e.g. painless lipohypertrophy, benign symmetric lipomatoses or lipomatosis dolorosa)
9. Other edema-causing diseases (such as lymphedema, phlebedema, or myxedema)
10. Lack of willingness to ensure adequate contraception
11. Positive pregnancy test
12. Breastfeeding
13. Use of a lymphomat
14. Participation in other clinical studies
15. Purely cosmetic reasons for participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lipedema is a symmetrical, congenital, excessive increase in fatty tissue on the legs, which occurs almost exclusively in women.
Enrollment: 450 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Successful Pain Reduction After 12 Months (≥ 2 Points on a Numeric Rating Scale) | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  The primary end point is the relevant reduction of the average pain of the last four weeks in the legs (≥ 2 points on a Numeric Rating Scale; German Pain Questionnaire) 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation.

SECONDARY OUTCOMES:
Change in Pain Severity as Assessed by German Pain Questionnaire | 12 months after completed liposuction treatment (intervention group) or after randomization (control group) compared with the time of randomisation)
  Change in severity according to von Korff et al. (1992) regarding pain in the legs (stage I, II or III). The severity is calculated based on the questions of the German Pain Questionnaire according to von Korff et al (1992). The assessment of the pain intensity as well as the impairment and information on the days of impairment are included in the calculation of the severity (classes 0 = no pain to 4 = high, pain-related impairment, strongly limiting).
Change in Health-Related Quality of Life According to SF-36 Questionnaire | 12 months after completed liposuction treatment (intervention group) or after randomization (control group) compared with the time of randomisation)
  Change in health-related quality of life according to SF-36 questionnaire.
Change in Health-Related Quality of Life According to DLQI Questionnaire | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Change in health-related quality of life according to DLQI questionnaire (a clinically relevant change corresponds to ≥ 4 points change in DLQI sum score).
Change in Health-Related Quality of Life According to WHOQOL-BREF Questionnaire | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Change in health-related quality of life according to WHOQOL-BREF questionnaire.
Change in Total Impairment According to Schmeller et al. (2010) | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Total impairment is measured by taking the mean of 7 numerical rating scales assessing the domains pain (spontaneous, pressure), swelling, hematoma, movement, cosmetic appearance and quality of life (0 (none) - 10 (always/very strong) points), see Schmeller et al. (2010).
Altered Depression Tendency According to PHQ-9 Questionnaire | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Altered depression tendency according to PHQ-9 questionnaire (a clinically relevant improvement corresponds to ≥ 5 points reduction in PHQ-9 sum score).
Altered Hematoma Tendency According to Schmeller et al. (2010) | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Hematoma ("Are you prone to bruising?") is measured by a numerical rating scale (0 (none) - 10 (always/very strong) points), see Schmeller et al. (2010).
Changed Prevalence of Edema | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Changed prevalence of edema
Change in the Scope of the Physical Therapy | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  The scope of the physical therapy is measured by the number of treatment sessions per month.
Change in Body Fat Percentage According to Wright et al. (1981) | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Change in body fat percentage, determined according to formula from Wright et al. (1981), collected by means of measuring tape at the following points:
  * abdominal circumference: measurement at the level of the navel. The tape measure is placed horizontally around the body
  * neck circumference: measurement below the larynx
  * body size
  * hip circumference: the widest part of the hip is measured.
Change of Leg Circumference by Means of Measuring Tape | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Change of leg circumference of the left and right leg by means of measuring tape at five specified measuring points:
  * lower leg cuffs
  * calf center
  * knee
  * 10 cm below the groin
  * hips (iliac crest).
Movement Restriction Reduction According to LEFS Sum Score | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Relevant reduction in movement restriction (stage I, II, or III; ≥ 9 points improvement in LEFS sum score)
Number of Recurrent Interventions | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Number of recurrent interventions
Number of (Serious) Adverse Events | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Number of (serious) adverse events
Number of Therapy Interruptions Caused by Adverse Events | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Discontinuation of therapy caused by adverse events
Optional: Change of the Leg Volume by Means of Perometry | 12 months after completed liposuction treatment (intervention group) or after randomisation (control group) compared with the time of randomisation)
  Optional: Change of the leg volume of the left and right leg (e.g. by means of perometry etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Podda, Dr. med., Study Chair — Hautklink Darmstadt
Locations (12):
- Germany (12):
  - Praxis für Dermatologie, Dermatochirurgie und Phlebologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Venenzentrum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Klinikum Ernst von Bergmann, Potsdam, Brandenburg
  - Hautmedizin Bad Soden, Bad Soden am Taunus, Hesse
  - Hautklinik Darmstadt, Darmstadt, Hesse
  - Hautarztpraxis Mühltal, Mühltal, Hesse
  - Evangelisches Krankenhaus Oldenburg Klinik für Plastische, Ästhetische, Rekonstruktive und Handchirurgie, Oldenburg, Lower Saxony
  - Johanniter GmbH Waldkrankenhaus Bonn, Bonn, North Rhine-Westphalia
  - Klinik und Praxisklinik für Plastische Chirurgie, Cologne, North Rhine-Westphalia
  - MVZ Praxis, Cologne, North Rhine-Westphalia
  - MVZ Praxis Dr. Cornely Düsseldorf MVZ Corius Nordrhein GmbH, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Podda M, Kovacs M, Hellmich M, Roth R, Zarrouk M, Kraus D, Prinz-Langenohl R, Cornely OA. A randomised controlled multicentre investigator-blinded clinical trial comparing efficacy and safety of surgery versus complex physical decongestive therapy for lipedema (LIPLEG). Trials. 2021 Oct 30;22(1):758. doi: 10.1186/s13063-021-05727-2. PMID 34717741